CLINICAL TRIAL: NCT02421419
Title: Pain With Trigger Finger Injection: A Comparison of Steroid Alone Versus Steroid/Lidocaine Mixture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed; recruitment problems
Sponsor: Kenneth Taylor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Kenneth Taylor, M.D., Associate Professor, Orthopaedics, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB - 001858
Record Dates: First submitted 2015-04-07; First posted 2015-04-20 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Trigger Finger Disorder
Keywords: flexor tendon entrapment; snapping finger; trigger digits; trigger thumb
MeSH Terms: conditions — Trigger Finger Disorder | interventions — dexamethasone 21-phosphate; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Corticosteroid alone (CS) Group (Active Comparator): 1 cc dexamethasone sodium phosphate (4mg/ml) injectable
  Interventions: Drug: Dexamethasone Sodium Phosphate
- Corticosteroid/Lidocaine (CSL) Group (Active Comparator): 1 cc dexamethasone sodium phosphate (4 mg/ml) injectable and 1 cc 1% Xylocaine (lidocaine) injectable
  Interventions: Drug: Dexamethasone Sodium Phosphate; Drug: Xylocaine
- Corticosteroid/Saline (CSS) Group (Active Comparator): 1 cc dexamethasone sodium phosphate (4mg/ml) injectable and 1 cc 0.9% injectable Sodium Chloride (saline)
  Interventions: Drug: Dexamethasone Sodium Phosphate; Drug: Sodium Chloride

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate — adreno-cortical steroid anti-inflammatory drug
  Other Names: Decadron phosphate
Drug: Xylocaine — a local anesthetic agent
  Other Names: Lidocaine HCL
  Arms: Corticosteroid/Lidocaine (CSL) Group
Drug: Sodium Chloride — Sodium chloride is a sterile, nonpryogenic solution for fluid and electrolyte replenishment
  Other Names: Saline
  Arms: Corticosteroid/Saline (CSS) Group

SUMMARY:
This research is being done to compare pain relief and efficacy of trigger finger injection using a combination of lidocaine/corticosteroid versus corticosteroid injection alone versus corticosteroid/saline combination.

DETAILED DESCRIPTION:
This is a prospective, randomized study comparing pain relief and efficacy of trigger finger injection using a combination of lidocaine/corticosteroid versus corticosteroid injection alone versus corticosteroid/saline combination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Male or female (non-pregnant)
* Clinically diagnosed trigger digit
* Subject is able to provide voluntary, written informed consent
* Subject, in the opinion of the clinical investigator, is able to understand the clinical investigation and is willing to perform all study procedures and follow-up visits.

Exclusion Criteria:

* Age <18 or >90
* Pregnant or lactating women
* Non-English speaking individuals
* Medication contradictions to lidocaine, corticosteroids and/or saline
* Prior injection or surgery on the affected finger
* Diagnosis of reflex symptomatic dystrophy (RSD) or complex regional pain syndrome (CRPS)
* Open wound

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Taylor, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saldana MJ. Trigger digits: diagnosis and treatment. J Am Acad Orthop Surg. 2001 Jul-Aug;9(4):246-52. doi: 10.5435/00124635-200107000-00004. PMID 11476534
- [Background] Strom L. Trigger finger in diabetes. J Med Soc N J. 1977 Nov;74(11):951-4. No abstract available. PMID 269967
- [Background] Kasdan ML, Leis VM, Lewis K, Kasdan AS. Trigger finger: not always work related. J Ky Med Assoc. 1996 Nov;94(11):498-9. PMID 8973080
- [Background] Marks MR, Gunther SF. Efficacy of cortisone injection in treatment of trigger fingers and thumbs. J Hand Surg Am. 1989 Jul;14(4):722-7. doi: 10.1016/0363-5023(89)90199-8. PMID 2754207
- [Background] Lambert MA, Morton RJ, Sloan JP. Controlled study of the use of local steroid injection in the treatment of trigger finger and thumb. J Hand Surg Br. 1992 Feb;17(1):69-70. doi: 10.1016/0266-7681(92)90014-s. PMID 1640148
- [Background] Murphy D, Failla JM, Koniuch MP. Steroid versus placebo injection for trigger finger. J Hand Surg Am. 1995 Jul;20(4):628-31. doi: 10.1016/S0363-5023(05)80280-1. PMID 7594291
- [Background] Maneerit J, Sriworakun C, Budhraja N, Nagavajara P. Trigger thumb: results of a prospective randomised study of percutaneous release with steroid injection versus steroid injection alone. J Hand Surg Br. 2003 Dec;28(6):586-9. doi: 10.1016/s0266-7681(03)00172-4. PMID 14599834

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
Started | 6 | 11 | 9
Completed | 6 | 11 | 8
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group | Total
Number analyzed (Participants) | 6 | 11 | 9 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 4 | 14
  >=65 years | 2 | 5 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 7 | 16
  Male | 5 | 3 | 2 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 11 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: VAS
Description: Visual Analogue Pain Scale (VAS) - measurement of pain on scale of 0 (least) to 10 (worst).
Time Frame: Patients are assessed pre-injection (baseline), 1 minute post-injection, 10 minutes post-injection, at 6 weeks post-injection and also asked to recollect their pain at time of injection when seen at 6 weeks post-injection
Population: VAS was collected on all study participants except for the one patient (CSS group) who was withdrawn after enrollment and before any measurements were taken.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
Number analyzed (Participants) | 6 | 11 | 8
units on a scale
  VAS pre-injection | 2.2 (1.0) | 3.0 (2.5) | 3.9 (2.9)
  VAS 1 minute post-injection | 2.3 (1.2) | 2.2 (2.6) | 4.9 (3.4)
  VAS 10 minutes post-injection | 2.1 (2.3) | 1.2 (1.7) | 3.3 (2.8)
  VAS 6 weeks post-injection | 1.5 (1.6) | 3.3 (3.7) | 4.0 (3.8)
  VAS Recollection | 5.2 (2.3) | 6.6 (2.5) | 5.9 (3.6)

2. Secondary Outcome: Presence of Triggering
Description: Patients are asked how often their finger triggers - not at all, rarely, occasionally, or frequently at time intervals indicated in the outcome measure time frame. Count of participants for each of these answers was collected.
Time Frame: Patients are assessed pre-injection (baseline), 1 minute post-injection, 10 minutes post-injection, and 6 weeks post-injection
Population: All participants from three groups were asked this question. Data was not collected on subject (CSS group) that withdrew from study after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
Number analyzed (Participants) | 6 | 11 | 8
Participants
  Triggering frequently pre-injection | 2 | 7 | 5
  Triggering not at all pre-injection | 0 | 0 | 2
  Triggering occasionally pre-injection | 4 | 4 | 1
  Triggering rarely pre-injection | 0 | 0 | 0
  Triggering not at all 1 minute post-injection | 3 | 1 | 3
  Triggering rarely 1 minute post-injection | 0 | 0 | 0
  Triggering occasionally 1 minute post-injection | 1 | 1 | 0
  Triggering frequently 1 minute post-injection | 0 | 0 | 0
  Triggering same as before 1 minute post-injection | 2 | 8 | 5
  Triggering not at all 10 minutes post-injection | 4 | 2 | 4
  Triggering rarely 10 minutes post-injection | 0 | 0 | 0
  Triggering occasionally 10 minutes post-injection | 1 | 1 | 0
  Triggering frequently 10 minutes post-injection | 0 | 1 | 0
  Triggering same as before 10 min. post-injection | 1 | 6 | 4
  Triggering not at all 6 wks post-injection | 3 | 1 | 1
  Triggering rarely 6 wks post-injection | 0 | 1 | 0
  Triggering occasionally 6 weeks post-injection | 0 | 0 | 0
  Triggering frequently 6 wks post-injection | 1 | 1 | 2
  triggering same as before 6 wks post-injection | 2 | 8 | 5

3. Secondary Outcome: Degree of Triggering
Description: A Green classification number (0-4) is given to each subject pre-injection and at 6 weeks post-injection based on their degree of triggering. 0 = No triggering, no pain; 1 = Pre-triggering; pain, history of catching, but not demonstrable on physical examination; tenderness over the A1 pulley; 2 = Active; demonstrable catching, but the patient can actively extend the digit; 3= Passive; demonstrable catching requiring passive extension or inability to actively flex; and 4 = Contracture; demonstrable catching with a fixed flexion contracture of the PIP joint.
Time Frame: Patients are assessed pre-injection objectively by investigator and at 6 weeks post-injection subjectively via Patient Survey
Population: Data collected on all subjects enrolled except for one that was withdrawn after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
Number analyzed (Participants) | 6 | 11 | 8
Participants
  Green classification 0 (pre-injection) | 0 | 0 | 0
  Green classification 1 (pre-injection) | 2 | 1 | 1
  Green classification 2 (pre-injection) | 4 | 10 | 6
  Green classification 3 (pre-injection) | 0 | 0 | 0
  Green Classification 4 (pre-injection) | 0 | 0 | 1
  Green classification 0 (6-weeks post-injection) | 2 | 1 | 1
  Green classification 1 (6-weeks post-injection) | 0 | 0 | 0
  Green classification 2 (6-weeks post-injection) | 2 | 2 | 4
  Green classification 3 (6-weeks post-injection) | 2 | 7 | 2
  Green classification 4 (6-weeks post-injection) | 0 | 1 | 1

4. Secondary Outcome: Number of Participants With Adverse Effects
Description: Incidence of adverse effects
Time Frame: Patients are assessed 1 minute post-injection, 10 minutes post-injection, and at 6 week post-injection.
Population: Adverse effects was collected on all study participants except for the one patient who was withdrawn after enrollment (CSS group)
Measure: Count of Participants; unit: Participants
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
Number analyzed (Participants) | 6 | 11 | 8
Participants
  Adverse effects 1 minute post-injection | 0 | 0 | 0
  Adverse effects 10 minutes post-injection | 0 | 0 | 0
  Adverse effects 6 weeks post-injection | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse effects were assessed 1 minute, 10 minutes, and 6 weeks post-injction
Arm/Group | Corticosteroid Alone (CS) Group | Corticosteroid/Lidocaine (CSL) Group | Corticosteroid/Saline (CSS) Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/8

LIMITATIONS AND CAVEATS:
Study closed prematurely on 1/25/2017 with 26 patients enrolled and 1 withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02421419/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02421419/ICF_001.pdf